CLINICAL TRIAL: NCT00160290
Title: An Open, Randomized, Parallel Group, Single Center Study to Investigate the Effect of Lactulose Versus Plantago Ovate on the Quality of Life of Patients With Hard Stools and Hemorrhoids or Anal Fissure
Brief Title: Trial to Evaluate Effect of Lactulose on Hard Stools in Patients With Hemorrhoids or Anal Fissures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This trial discontinued on 30 JUN 2006 due to a lack of enrolment
Sponsor: Solvay Pharmaceuticals (Industry)
Responsible Party: David Vilardell, Solvay Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S105.4.106
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-04

CONDITIONS: Hemorrhoids; Anal Fissures
Keywords: lactulose; randomised clinical trial; hemorrhoids; anal fissures
MeSH Terms: conditions — Hemorrhoids; Fissure in Ano | interventions — Lactulose; Psyllium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Lactulose Group
  Interventions: Drug: Lactulose
- B (Active Comparator): Plantago Group
  Interventions: Drug: Plantago ovata

INTERVENTIONS:
Drug: Lactulose — 15 mL / 12 hours
  Arms: A
Drug: Plantago ovata — 3,5 g / 12 hours
  Arms: B

SUMMARY:
To demonstrate that lactulose acts as a stool softener, relieving the pain at defecation, improving the number of defecations and regulating the colonic transit time in patients suffering of hemorrhoids or anal fissure. To compare efficacy and quality of life in patients treated either with lactulose or plantago ovate.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from symptomatic hemorrhoids, or symptomatic anal fissure.

Exclusion Criteria:

* Patients suffering from malignant tumor in the intestine or the anal-rectal region, irritable colon, intestine inflammatory disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2002-03; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Quality of life of patients with hard stools and hemorrhoids or anal fissure | 6 weeks

SECONDARY OUTCOMES:
Gastrointestinal Symptoms Rating Scale | 6 weeks
Bristol stool consistency scale | 6 weeks
Number of episodes of rectal bleeding | 6 weeks
Need of rescue medication | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (8):
- Spain (8):
  - Site 2, Barcelona
  - Site 6, Granada
  - Site 5, Huesca
  - Site 7, Oviedo
  - Site 4, Sabadell (Barcelona)
  - Site 3, Sant Cugat Del Vallès (Barcelona)
  - Site 8, Santiago de Compostela
  - Site 1, Valencia